CLINICAL TRIAL: NCT05249114
Title: Phase Ib Study of Cabozantinib in Combination With Lu-177 DOTATATE Peptide Receptor Radionuclide Therapy (PRRT) in Patients With Progressive, Previously Treated Somatostatin Receptor 2 (SSTR2) Positive Neuroendocrine Tumors (NETs)
Brief Title: Study of Cabozantinib With Lu-177 in Patients With Somatostatin Receptor 2 Positive Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Exelixis (Industry); Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022000050
Record Dates: First submitted 2022-01-31; First posted 2022-02-21 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Neuroendocrine Tumors
Keywords: Phase 1b; Cabozantinib; Lu-177; Lutathera; SSTR2; Gastrointestinal
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — cabozantinib; Lutetium-177; lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1 (Experimental): Cabozantinib 20 mg daily with Lu-177 DOTATE administration IV. For cycles 5+, single-agent maintenance of cabozantinib is given at 20 mg qd.
  Interventions: Drug: Cabozantinib; Drug: Lu-177
- Cohort 2 (Experimental): Cabozantinib 40 mg qod alternating with 20 mg qod with Lu-177 DOTATE administration IV. For cycles 5+, single-agent maintenance of cabozantinib is given at 40 mg qd.
  Interventions: Drug: Cabozantinib; Drug: Lu-177
- Cohort 3 (Experimental): Cabozantinib 40 mg qd with Lu-177 DOTATE administration IV. For cycles 5+, single-agent maintenance of cabozantinib is given at 40 mg qd.
  Interventions: Drug: Cabozantinib; Drug: Lu-177
- Cohort 4 (Experimental): Cabozantinib 60 mg qod alternating with 40 mg qod with Lu-177 DOTATE administration IV. For cycles 5+, single-agent maintenance of cabozantinib is given at 60 mg qd.
  Interventions: Drug: Cabozantinib; Drug: Lu-177
- Cohort 5 (Experimental): Cabozantinib 60 mg qd with Lu-177 DOTATE administration IV. For cycles 5+, single-agent maintenance of cabozantinib is given at 60 mg qd until disease progression.
  Interventions: Drug: Cabozantinib; Drug: Lu-177

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib tablets are supplied as film coated tablets containing cabozantinib malate equivalent to 20 mg and 60 mg of cabozantinib and contain microcrystalline cellulose, lactose anhydrous, hydoxypropyl cellulose, croscarmellose sodium, colloidal silicon dioxide, magnesium stearate and Opadry yellow. The 60 mg tablets are oval and the 20 mg tablets are round. Doses of 40 mg will comprise two 20-mg tablets.
  Other Names: Cabometyx
Drug: Lu-177 — Currently, the only FDA-approved PRRT consists of dotatate, a somatostatin analogue, radiolabeled with Lutetium-177 (Lu177), a beta-minus emitter (brand name Lutathera). Lu177 induces cell death via DNA strand breaks, caspase-3 apoptosis, and interfering with DNA-PK expression (which is associated with DNA repair). PRRT with Lu-177 DOTATATE is a targeted, intravenous therapy inducing DNA damage by delivering ionizing radiation to somatostatin receptor positive tumors.
  Other Names: Lutathera

SUMMARY:
The phase I objective of this study is to establish the maximal tolerated dose (MTD) of cabozantinib in 20 mg, 40 mg and 60 mg dose escalation cohorts in combination with Lu-177 dotatate at a standard dose of 7.4 GBq in four (4) 8-week cycles followed by continuation cabozantinib.

DETAILED DESCRIPTION:
Patients will be treated four (4) cycles of combination cabozantinib with Lu-177 DOTATATE followed by maintenance cabozantinib. Cycles 1-4 combination cabozantinib with Lu-177 DOTATATE is given in 8-week cycles, with cabozantinib initiated on day 1 and Lu-177 DOTATATE given on day 14. Cabozantinib dosing is escalated during cycles 1-4 in the following manner: dose cohort 1 patients receive cabozantinib 20 mg daily, cohort 2 receive 40mg qod alternating with 20 mg qod, cohort 3 receive 40 mg qd, dose cohort 4 receive 60 mg qod alternating with 40 mg qod, and dose cohort 5 receive 60 mg qd. In all cohorts, during cycle 5 and beyond, single-agent maintenance cabozantinib is given in 4-week cycles in a qd dosing scheduling as follows: 20 mg qd cohort 1; 40 mg qd cohort 2; 40 mg qd cohort 3; 60 mg qd cohort 4; 60 mg qd cohort 5, until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unresectable, progressive, histologically well-differentiated neuroendocrine tumors of the fore-, mid-, or hindgut, including pancreas, or those with an unknown primary with target lesions overexpressing somatostatin receptors (Krenning 2, 3 or 4) on a SSTR PET.
2. Patients must have previously received one or more lines of systemic therapy including somatostatin analogue therapy.
3. Prior PRRT therapy is permitted up to a maximum of 4 standard doses. Enrollment of R-PRRT patients is permitted after initially 3 PRRT-naïve patients have been enrolled on protocol and if the minimum progression free survival (PFS) with initial PRRT therapy was ≥ 18 months from day 1, cycle 1 of PRRT to progression.
4. ECOG 0-2.
5. Recovery to baseline or ≤ Grade 1 (CTCAE v5.0) from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
6. Minimum 18 years or older.
7. Adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 14 days before first dose of study treatment:

   1. Absolute neutrophil count (ANC) ≥ 1500/µL without granulocyte colony-stimulating factor support.
   2. White blood cell count ≥ 2500/µL.
   3. Platelets ≥ 100,000/µL without transfusion.
   4. Hemoglobin ≥ 9 g/dL (≥ 90 g/L).
   5. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x upper limit of normal (ULN). ALP ≤ 5 x ULN with documented bone metastases.
   6. Total bilirubin ≤ 1.5 x ULN (for patients with Gilbert's disease ≤ 3 x ULN).
   7. Serum albumin ≥ 2.8 g/dl
   8. (PT)/INR or partial thromboplastin time (PTT) test < 1.3 x the laboratory ULN
   9. Serum creatinine ≤ 2.0 x ULN or estimated creatinine clearance ≥ 30 mL/min (≥ 0.5 mL/sec) using the Cockcroft-Gault equation:

      Males: (140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72) Females: [(140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)] × 0.85
   10. Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol), or 24-h urine protein ≤ 1 g
8. Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.
9. Sexually active fertile participants and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment.
10. Female participants of childbearing potential must not be pregnant at screening. Female participants are considered to be of childbearing potential unless one of the following criteria are met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating (FSH) level > 40 mIU/mL to confirm menopause). Note: Documentation may include review of medical records, medical examinations, or medical history interview by study site.

Exclusion Criteria:

1. Prior therapy with cabozantinib.
2. Tumors with poorly differentiated or small cell histology.
3. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
4. Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment.
5. Radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Participants with clinically relevant ongoing complications from prior radiation therapy are not eligible.
6. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis). Participants must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible participants must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment.
7. Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

   1. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
   2. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
8. The participant has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   a. Cardiovascular disorders: i. Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.

   ii. Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.

   iii. Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose of study treatment.
   1. Participants with a diagnosis of incidental, subsegmental PE or DVT within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation (see exclusion criterion #6) for at least 1 week before first dose of study treatment.
   2. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

   i. The participant has evidence of tumor invading into the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), active diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.

   ii. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment.

   iii. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.
9. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
10. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
11. Other clinically significant disorders that would preclude safe study participation.

    1. Serious non-healing wound/ulcer/bone fracture.
    2. Uncompensated/symptomatic hypothyroidism.
    3. Moderate to severe hepatic impairment (Child-Pugh B or C).
12. Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal or biopsy of brain metastasis) within 2 weeks before first dose of study treatment. Minor surgeries within 10 days before first dose of study treatment. Participants must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Participants with clinically relevant ongoing complications from prior surgery are not eligible.
13. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 14 days before first dose of study treatment [add reference for Fridericia formula].

    Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.
14. Pregnant or lactating females.
15. Inability to swallow tablets.
16. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
17. Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Establish the maximal tolerated dose of cabozantinib in combination with Lu-177 dotatae at a standard dose of 7.4 GBg in four 8-week cycles followed by continuation of cabozantinib. | Up to 2 years
  The phase I objective of this study is to establish the maximal tolerated dose (MTD) of cabozantinib in 20 mg, 40 mg and 60 mg dose escalation cohorts in combination with Lu-177 dotatate at a standard dose of 7.4 GBq in four (4) 8-week cycles followed by continuation cabozantinib. Due to overlapping toxicities of cabozantinib and Lu-177 dotatate and to allow more incremental dose escalation of cabozantinib, alternating day dosing of 40mg/20mg and 60mg/40mg cohorts are incorporated into the schema. This is expected to reduce the risk of overlapping toxicities while still achieving radio-sensitizing anti-angiogenic, multi-targeted therapy in combination with the beta-emitting radiation from lutetium 177 synergistic due to the prolonged half-life of cabozantinib.

SECONDARY OUTCOMES:
Establish objective response rate as measured by RECIST 1.1 | Up to 2 years post study completion
  The secondary outcome measure is to establish the objective response rate (ORR) as measured by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Imaging is done every 16 weeks and/or re-staging through study completion up to 2 years. A minimum observed overall response rate (ORR) of ≥ 25% in the PRRT-naïve cohort, as measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 in the treatment population would justify further randomized efficacy studies.

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Kennecke, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Cancer Institute - Franz Clinic, Portland, Oregon, United States